CLINICAL TRIAL: NCT05600517
Title: Evaluation of Caries Prevention Based on Genetic Etiology and Risk: Protocol for a Multicenter Randomized Controlled and Adaptive Trial for Oral Personalized Care (PRECARIES)
Brief Title: Evaluation of Caries Prevention Based on Genetic Etiology and Risk.
Acronym: PRECARIES
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Umeå University (Other)
Collaborators: Vastra Gotaland Region (Other Government); Region Västerbotten (Other Government); Region Skane (Other); Region Halland (Other); Uppsala-Örebro Regional Research Council (Other); Region Östergötland (Other); Region Gävleborg (Other); County Council of Norrbotten, Sweden (Other Government); Västernorrland County Council, Sweden (Other Government); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Dnr 2020-02533
Record Dates: First submitted 2022-10-20; First posted 2022-10-31 (Actual); Last update posted 2022-10-31 (Actual); Status verified 2022-10

CONDITIONS: Caries,Dental
Keywords: caries; genetic; prevention; saliva; S. Mutans; lifestyle; microbiota; exposure; Proline rich protein gene 1 (PRH1); Proline rich protein gene 2 (PRH2); Deleted malignant brain tumour (DMBT-1)
MeSH Terms: conditions — Dental Caries | interventions — Fluorides

STUDY DESIGN:
Intervention Model Description: Randomized controlled study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Participant is not informed about if they are in the control or intervention group Outcome assessor are not aware of group allocation Both dentist/nurse and patient do not know the genotype or risk group. Caries registration at start and end will be performed by a dentist not involved in giving the orthodontic treatment or prevention to each patient
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Standard prevention fluoride P4+ (No Intervention): self-care prevention on diet, oral hygiene and fluoridated toothpaste 1450 ppm with checkup every second month with one occasion of fluoride varnish at the clinic.
- Intensive prevention P4+ (Experimental): a patient-centered education on diet, oral hygiene and fluoridated toothpaste 5000ppm with check up´s and topical fluoride application (varnish) every second month.
  Interventions: Other: Fluoride
- Standard prevention fluoride P4- (No Intervention): self-care prevention on diet, oral hygiene and fluoridated toothpaste 1450 ppm with checkup every second month with one occasion of fluoride varnish at the clinic.
- Intensive prevention P4- (Experimental): a patient-centered education on diet, oral hygiene and fluoridated toothpaste 5000ppm with check up´s and topical fluoride application (varnish) every second month.
  Interventions: Other: Fluoride

INTERVENTIONS:
Other: Fluoride — a patient-centered education on diet, oral hygiene and fluoridated toothpaste 5000ppm with check up´s and topical fluoride application (varnish) every second month.
  Arms: Intensive prevention P4+; Intensive prevention P4-

SUMMARY:
Dental caries affects billions of people worldwide and involves saliva immunodeficiency, commensal pathogen and exposure (lifestyle) causal subtypes of the disease. Up to 85% of adolescents in Swedish and other low prevalence populations are caries-free while the remaining 15% show high, recurrent caries activity. Accordingly, there is a lack of cost-effective risk assessment and prevention tools for personalized oral care. This randomized adaptive clinical trial (RCT) evaluates both caries prevention based on genetic etiology and risk, as a consequence of saliva immunodeficiency genes specifying individuals as susceptible or resistant to caries, and the effect of intensified versus selfcare traditional prevention on the two groups.

DETAILED DESCRIPTION:
This is a protocol for a multicenter risk assessment and intervention study (PRECARIES) with an adaptive component. The study design comprises a prescreen of 2000 adolescents of which 520 will be included in the RCT study part with adolescents undergoing ordinary orthodontic treatment with multibrackets at the Public Dental Service. The orthodontic treatment allows for rapid caries development and improved discrimination between susceptible versus resistant individuals. The children are genotyped into two risk groups; genetic susceptible and non-susceptible children that are assigned to intensive or traditional standard prevention. The clinical outcomes will adaptively be measured at different time points (0, 6, 12 and months) as caries lesions at different teeth and surfaces using tactile, visual and X-ray bitewing, clinical photos and quantitative laser fluorescence (QLF). Secondary outcomes will be inflammation at the gingival margins and pocket depth at debonding of the orthodontic appliances. Questionaires are collected as well as biological samples; swab-dna, whole and parotid saliva and microbiota. Human and microbiota geno-and protein typing involves in and ex house platforms adaptively.

ELIGIBILITY:
Inclusion Criteria:

- undergoing orthodontic treatment with fixed multibrackets appliance in the upper and lower arch

Exclusion Criteria:

* impacted canines
* agenesis in the frontal region
* maxillofacial surgery

Ages: 13 Years to 23 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 520 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-01-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
% change in increment DeFS (decayed, enamel included and filled tooth surfaces) | 6 months
  The % change in ΔDeFS caries increment over a follow up period of 6 and 24 months related to prevention.
% change in increment DeFS (decayed, enamel included and filled tooth surfaces) | 24 months
  The % change in ΔDeFS caries increment over a follow up period of 6 and 24 months related to prevention.
DFS (decayed and filled tooth surfaces) and DeFS (decayed, enamel included and filled tooth surfaces) | Baseline (0 months)
  The baseline and prospective caries scores for incidence and progression of lesions related to risk group
DFS (decayed and filled tooth surfaces) and DeFS (decayed, enamel included and filled tooth surfaces) | 6 months
  The baseline and prospective caries scores for incidence and progression of lesions related to risk group
DFS (decayed and filled tooth surfaces) and DeFS (decayed, enamel included and filled tooth surfaces) | 24 months
  The baseline and prospective caries scores for incidence and progression of lesions related to risk group

SECONDARY OUTCOMES:
Gingival inflammation | Baseline (0 months)
  Bleeding on probing quadrant 3, Gingival inflammation will be represented by the index Bleeding on probing (BoP). BoP will be performed at the buccal surfaces in the third quadrant of the mouth approximately 21 surfaces
Gingival inflammation | 6 months
  Bleeding on probing quadrant 3, Gingival inflammation will be represented by the index Bleeding on probing (BoP). BoP will be performed at the buccal surfaces in the third quadrant of the mouth approximately 21 surfaces
Gingival inflammation | 24 months
  Bleeding on probing quadrant 3, Gingival inflammation will be represented by the index Bleeding on probing (BoP). BoP will be performed at the buccal surfaces in the third quadrant of the mouth approximately 21 surfaces
Mineralization disorders | Baseline (0 months)
  Mineralization disturbances in enamel, including fluorosis, molar-incisor-hypo-mineralization, amelogenesis imperfecta are noted in the clinical examinations and by viewing clinical photographs and QLF technique.
Mineralization disorders | 6 months
  Mineralization disturbances in enamel, including fluorosis, molar-incisor-hypo-mineralization, amelogenesis imperfecta are noted in the clinical examinations and by viewing clinical photographs and QLF technique.
Mineralization disorders | 24 months
  Mineralization disturbances in enamel, including fluorosis, molar-incisor-hypo-mineralization, amelogenesis imperfecta are noted in the clinical examinations and by viewing clinical photographs and QLF technique.

OTHER OUTCOMES:
Life style variables | Baseline (0 months)
  Sociodemographic data (sex and ethnicity), oral hygiene, intake frequency of sweets (e.g., cookies, biscuits, ice cream or dried fruit) and sugary drinks (never, once per month, once per week, several times per week, once per day, several times per day), and the use of extra fluoride
Life style variables | 24 months
  Sociodemographic data (sex and ethnicity), oral hygiene, intake frequency of sweets (e.g., cookies, biscuits, ice cream or dried fruit) and sugary drinks (never, once per month, once per week, several times per week, once per day, several times per day), and the use of extra fluoride
Microbiota | Baseline (0 months)
  Number and type of S. mutans
Microbiota | 24 months
  Number and type of S. mutans

CONTACTS AND LOCATIONS:
Overall Officials: Nicklas Stromberg, Prof, Principal Investigator — Umeå University
Locations (1):
- Umeå University Hospital, Umeå, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stromberg N, Esberg A, Sheng N, Marell L, Lofgren-Burstrom A, Danielsson K, Kallestal C. Genetic- and Lifestyle-dependent Dental Caries Defined by the Acidic Proline-rich Protein Genes PRH1 and PRH2. EBioMedicine. 2017 Dec;26:38-46. doi: 10.1016/j.ebiom.2017.11.019. Epub 2017 Nov 22. PMID 29191562
- See also: E Biomedicine publication — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5832611/
- Available data/document: Clinical Study Report: 10.1016/j.ebiom.2017.11.019 — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5832611/